CLINICAL TRIAL: NCT01112930
Title: n-3 Fatty Acids and Early Child Nutrition: 5-Year-Olds X-Section Study
Brief Title: Essential Fatty Acid (EFA) Nutrition 5-Year-Olds X Section
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: H09-02921
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Breastfeeding
Keywords: essential fatty acids; DHA; preschool children; docosahexanoic acid (DHA)
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma and blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
In humans, docosahexanoic acid (DHA) is concentrated in brain. After birth, DHA is obtained from breast milk or the child's diet. The investigators are studying whether DHA intakes in young children are adequate to support brain development. This is a cross-sectional study of children 5-6 years-old.

DETAILED DESCRIPTION:
This research involves recruitment of a cross-sectional cohort of children 5 years of age and their mothers. The purpose is to assess the relationship between the child's diet, DHA status and neural, cognitive and behavioral development. Hypotheses: 1. Children with low DHA status will be at increased risk for poor scores on tests of development. 2. Family food practices will be major determinant of DHA intake of preschool children in our population. 3. Genetic variation in fatty acid metabolism will influence blood fatty acids in preschool children.

Objectives: 1. To determine if low DHA status among children 5-6 years-of-age is associated with low scores on tests of development; 2. To identify the dietary patterns that place children at risk for poor DHA status, 3. To show genetic variation also alters blood fatty acids in children.

This research will recruit a cohort of 5-6year-old children (n= 200). Subjects will attend our nutrition lab at the Child and Family Research Institute where the child will complete play-like developmental assessments. Measurement of blood pressure, heart rate, height and weight will be completed and blood samples will be collected to measure DHA status and polymorphisms (SNP) in genes of fatty acid metabolism. The parent will be asked to provide information on the child' diet and health. Baseline characteristics for the subjects will be summarized using descriptive statistics. Logistic regression will be used to assess the relationship of DHA status to cognitive development with multi-variable-adjusted odds ratios (ORs) of a negative outcome and corresponding 95% confidence interval (CI). Regressions will also be run with the outcomes in continuous form to assess the changes in scores associated with increments of child DHA status. For all multivariate regression models, potential confounders will be screened in stepwise fashion, and any covariate with a regression coefficient P-value < 0.05 (two-sided) will be retained. Variables will include gender, birth weight, gestation length, maternal intelligence quotient (IQ), ethnicity, breast-feeding duration, birth order, and dichotomized variables of child health, eating behavior and martial status. Children will grouped in quintiles of blood DHA and descriptive statistics will be used to present intakes of total fat, individual fatty acids. ANOVA will be used to determine if genetic variables in Fetal Akinesia Deformation Sequence (FADS) influence blood DHA.

ELIGIBILITY:
Inclusion Criteria:

* comfortable to speak and read in English
* parent or primary caregiver of a healthy child that is 5-6 years of age.

Exclusion Criteria:

* not capable/comfortable with reading, speaking and writing the English language.
* not the parent or primary caregiver or legal guardian of a 5-6 year-old child.
* the child that is not in good health or has severe food allergies or a metabolic, neurological, genetic, or immune disorder that influences the child's food choices will not be able to participate in this study.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This is a cross-sectional study of children 5-6 years-old.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
plasma lutein and red blood cell DHA | 5 years 8 months to 6 years
  plasma lutein and red blood cell DHA biochemistries

SECONDARY OUTCOMES:
cognitive development with standardized developmental tests | 5 years 8 months to 6 years
  Assessment with the Kaufman Developmental Assessment Battery

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Dr., Principal Investigator — University of British Columbia; Tim Oberlander, MD, Study Director — University of British Columbia
Locations (1):
- Child & Family Research Institute, Nutrition and Metabolism Research Program, Vancouver, British Columbia, Canada